CLINICAL TRIAL: NCT04334889
Title: Differences in Spinal Kinematics During Various Activities Between Asymptomatic Subjects and Patients With Chronic Low Back Pain
Brief Title: Measurement of Spinal Kinematics During Various Movements
Status: Not yet recruiting | Type: Observational
Sponsor: Haute Ecole de Santé Vaud (Other)
Collaborators: University of Lausanne Hospitals (Other); Clinique Romande de Readaptation (Network)
Responsible Party: Sponsor
Other Study IDs: LBP2020
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic low back pain (CLBP): All CLBP patients should present with non-specific low back pain (pain from lower ribs to gluteal folds) for more than 3 months.
  Interventions: Other: Visual cues
- Asymptomatic controls: Asymptomatic participants should have had no history of LBP requiring medical attention during the last two years and no other concomitant pain or condition that could compromise the evaluation of lumbar kinematics.
  Interventions: Other: Visual cues

INTERVENTIONS:
Other: Visual cues — Participants will be asked to move following cues displayed on a screen in front of them.

SUMMARY:
Participants will perform movements while receiving different visual cues. Spinal kinematics will be measured during these movements and compared between asymptomatic and CLBP participants. Participants will come for a unique session.

ELIGIBILITY:
Inclusion Criteria:

- sufficient French level to understand the instructions for the tests, the information sheet, the consent form.

For CLBP patients:

- diagnosis of non-specific low back pain (pain from lower ribs to gluteal folds) for more than 3 months.

For asymptomatic participants:

* no history of LBP requiring medical attention during the last two years
* no other concomitant pain or condition that could compromise the evaluation of lumbar kinematics.

Exclusion Criteria:

* pregnancy
* skin allergy to tape
* body mass index (BMI) above 32

For patients with CLBP only:

* specific low back pain (such as the presence of infection, rheumatological or neurological diseases, spinal fractures, tumours)
* any known important spinal deformities
* previous back surgery that limits spinal mobility
* high level of pain at the time of experiment that prevents repeated movements (severity and irritability)
* other concomitant pain or condition that could compromise the evaluation of spinal kinematics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CLBP patients will be recruited through a multimodal rehabilitation program at Lausanne University Hospital, medical doctors or physiotherapists' consultations.
  Healthy controls will be a convenience sample recruited using flyers and emails, notably posted at the Lausanne University Hospital, the University of Health Professions in Lausanne (HESAV) and at the University of Lausanne.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Spinal kinematics | Day 1
  Spinal kinematics will be measured at the lumbar and thoracic spine in degrees

IPD SHARING:
Plan to Share IPD: No